CLINICAL TRIAL: NCT06765941
Title: Clinical Validation of Probe-based Parathyroid Autofluorescence Detection System PTeye vs Surgeons Eyes in Intraoperative Identification and Functional Preservation of Parathyroid Glands During Thyroid Surgery: A Parallel Randomized Controlled Clinical Trial.
Brief Title: PTeye vs Surgeons Eyes in Intraoperative Identification and Functional Preservation of Parathyroid Glands During Thyroid Surgery: A Parallel Randomized Controlled Clinical Trial.
Acronym: PTSURGEYE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marcin Barczynski (Other)
Responsible Party: Sponsor-Investigator, Marcin Barczynski, Head, Department of Endocrine Surgery, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N41/DBS/001474
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Surgery; Parathyroid Dysfunction; Hypoparathyroidism Post-surgical
Keywords: thyroid surgery; postoperative hypoparathyroidism; near-infrared autofluorescence; PTeye; probe-based parathyroid detection; visual identification
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thyroid operations with PTeye system for parathyroid glands identification (Experimental)
  Interventions: Device: Probe-based near-infrared parathyroid autofluorescence detection system
- Thyroid operations with surgeons naked eyes for parathyroid glands identification without PTeye (Active Comparator)
  Interventions: Procedure: Surgeons naked eyes for parathyroid glands identification

INTERVENTIONS:
Device: Probe-based near-infrared parathyroid autofluorescence detection system — The surgeon will use the PTeye as an intraoperative tool to identify whether a suspect tissue is parathyroid or not during the surgery. The surgeon will first take five baseline NIRAF measurements on the thyroid gland (or neck muscle, if thyroid is absent), to establish a reference point for subsequent measurements, using the disposable sterile fiber probe that is connected to the PTeye console, as per device functionality requirements. The subsequent step involves touching the target tissue in the neck with the fiber optic probe, after which the PTeye will indicate to the surgeon whether the tissue is parathyroid or not. Parameters displayed on the PTeye console - Baseline values, Detection Intensity, Parathyroid Detection Ratio - will be recorded for each patient in the study arm. PTeye indicates that a tissue is parathyroid if the 'Parathyroid Detection Ratio' is greater than 1.2. The rest of the surgical procedure will follow the standard protocol.
  Arms: Thyroid operations with PTeye system for parathyroid glands identification
Procedure: Surgeons naked eyes for parathyroid glands identification — The surgeons will not use the probe-based near-infrared parathyroid autofluorescence detection system and will proceed with the procedure as usual, relying on their surgical experience to identify parathyroid glands. At the end of the procedure, the thyroid specimen will be evaluated visually to search for inadvertently resected parathyroid glands. If this is the case, these parathyroid glands will be reimplanted in the sternocleidomastoid muscle, following standard protocol.
  Arms: Thyroid operations with surgeons naked eyes for parathyroid glands identification without PTeye

SUMMARY:
The goal of this randomized clinical trial is to learn if there are any added benefits of using near-infrared autofluorescence (NIRAF) probe-based imaging system (the PTeye) for intraoperative identification of parathyroid glands (PGs) during thyroid surgery in comparison to visual identification of PGs by the surgeon's naked eyes without PTeye.

The main questions it aims to answer are:

* Is number of PGs identified intraoperatively and preserved in situ larger in thyroid operations with PTeye versus surgeon's naked eyes without PTeye?
* Is number of patients with undetectable or low parathormone serum level on postoperative day 1 fewer in thyroid operations with PTeye versus surgeon's naked eyes without PTeye?
* Is number of patients requiring substitution therapy with calcium and vitamin D analogue fewer after thyroid operations with PTeye versus surgeon's naked eyes without PTeye in a short-term (< 6 weeks) and/or in a long-term (at 6 months) follow-up?
* Is numer of inadvertenly removed and reimplanted PGs fewer in thyroid operations with PTeye versus surgeon's naked eyes without PTeye?
* Is number of frozen sections fewer in thyroid operations with PTeye versus surgeon's naked eyes without PTeye?
* Is number of PGs identified by pathologist in the surgical specimen fewer in in thyroid operations with PTeye versus surgeon's naked eyes without PTeye?
* Is number of patients with symptomatic hypoparathyroidism within 30 days of the operation fewer in thyroid operations with PTeye versus surgeon's naked eyes without PTeye? The hypothesis explored in this study is that use of PTeye in comparison to the surgeon's naked eyes may be beneficial for intraoperative identification and preservation of PGs in thyroid surgery leading to reduced risk of postoperative hypoparathyroidism.

A prospective, randomized study with 2 arms: use of PTeye vs. visual identification of PGs without PTeye (n=77 patients, each).

The primary outcome measure is number of intraoperatively identified PGs with use of PTeye vs without it.

DETAILED DESCRIPTION:
A single-center prospective study with 1:1 randomization and a control group. It was assumed that it is possible to visually identify 2-3 (average 2.5) out of 4 PGs (62.5%), and that the use of the PTeye probe will increase the number of identified PGs to 3-4 (average 3.5) out of 4 (87, 5%). The statistical power for p<0.05 and 90% sensitivity of the study designed in this way is 122 patients (61 in each group), and taking into account the 20% risk of patients withdrawal or dropping out from the study, the required number is 154 patients, 77 patients in each group.

Inclusion criterion: a patient with thyroid disease qualified for first-time total thyroidectomy.

Exclusion criteria: history of thyroid or parathyroid surgery, planned simultaneous thyroid and parathyroid surgery, renal failure, pregnancy, lactation, allergy to contrast agents and/or iodine, inability of the patient to understand the study protocol, inability to participate in the planned postoperative follow-up, age below 18 years.

Included patients will be randomly assigned to the study group (thyroid surgery with the PTeye device) or the control group (thyroid surgery without the device).

Randomization will be performed on the Eurocrine platform. The PTeye device will be used in the study group for intraoperative identification of the PGs. In the control group, the PGs will be identified using the classic technique based on visual identification with naked eyes.

For patients assigned to the study arm with PTeye:

The surgeon will use the PTeye as an intraoperative tool to identify whether a suspect tissue is parathyroid or not during the surgery. The surgeon will first take five baseline NIRAF measurements on the thyroid gland (or neck muscle, if thyroid is absent), to establish a reference point for subsequent measurements, using the disposable sterile fiber probe that is connected to the PTeye console, as per device functionality requirements. The subsequent step involves touching the target tissue in the neck with the fiber optic probe, after which the PTeye will indicate to the surgeon whether the tissue is parathyroid or not. Parameters displayed on the PTeye console - Baseline values, Detection Intensity, Parathyroid Detection Ratio - will be recorded for each patient in the study arm. PTeye indicates that a tissue is parathyroid if the 'Parathyroid Detection Ratio' is greater than 1.2. The rest of the surgical procedure will follow the standard protocol. At the end of the procedure, the thyroid specimen will be evaluated with the PTeye to search for inadvertently resected parathyroid glands. If found, these parathyroid glands will be reimplanted in the sternocleidomastoid muscle, following standard protocol.

For patients assigned to the control arm without PTeye:

The surgeon will not use the PTeye and will proceed with the procedure as usual, relying on their surgical experience to identify parathyroid glands. At the end of the procedure, the thyroid specimen will be evaluated visually to search for inadvertently resected parathyroid glands. If this is the case, these parathyroid glands will be reimplanted in the sternocleidomastoid muscle, following standard protocol.

Preoperative, intraoperative, and postoperative parameters measured for all patients:

The following data will be compiled for all enrolled patient: patient demographics, duration of surgery, number of frozen section analyses performed, frozen section and permanent histology reports of all excised tissues, blood calcium levels (before surgery, on 1st post-operative day, on 1st postoperative visit after surgery, and at 6 months after surgery (if followed up)), parathyroid hormone (PTH) serum levels (on 1st post-operative day, on 1st postoperative visit after surgery, and at 6 months after surgery (if followed up)), history and duration of calcium and/or Vitamin D supplementation before and after surgery, and postsurgical complications, if any, and history of emergency room visits or hospitalization.

These preoperative, intraoperative, and postoperative investigations will be performed at the surgeon's discretion as necessary for the patient and as standard management for patients with thyroid pathologies. These parameters will then be compared between the study arm and the control arm to gauge the impact or value of PTeye suystem for thyroid surgeries.

ELIGIBILITY:
Inclusion Criteria:

* a patient with thyroid disease qualified for first-time total thyroidectomy.

Exclusion Criteria:

* history of thyroid or parathyroid surgery,
* planned simultaneous thyroid and parathyroid surgery,
* renal failure,
* pregnancy,
* lactation,
* allergy to contrast agents and/or iodine,
* inability of the patient to understand the study protocol,
* inability to participate in the planned postoperative follow-up,
* age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of intraoperatively identified parathyroid glands | During thyroid operation

SECONDARY OUTCOMES:
Numer of inadvertenly removed and reimplanted parathyroid glands | During thyroid surgery
Number of frozen sections | During thyroid surgery
Numer of patients with undetectable or low parathormone serum level | Postoperative day 1
Number of parathyroid glands identified by pathologist in the surgical specimen | Within 30 days postoperatively
Number of patients requiring substitution therapy with calcium and vitamin D analogue | At 30 days postoperatively
Number of patients with symptomatic hypoparathyroidism | Within 30 days postoperatively
Number of patients requiring substitution therapy with calcium and vitamin D analogue | At 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrine Surgery, Faculty of Medicine, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abood A, Rolighed L, Ovesen T, Madsen SH, Vestergaard P, Triponez F. Autofluorescence-guided hemithyroidectomy in a low-volume thyroid institution with no experience in parathyroid surgery: randomized clinical trial. Br J Surg. 2024 Apr 3;111(4):znae075. doi: 10.1093/bjs/znae075. PMID 38573333
- [Background] Vetter D, Triponez F. Near-infrared fluorescence techniques to reduce hypocalcaemia after thyroidectomy. Br J Surg. 2023 Nov 9;110(12):1590-1593. doi: 10.1093/bjs/znad221. No abstract available. PMID 37463423
- [Background] Vidal Fortuny J, Belfontali V, Sadowski SM, Karenovics W, Guigard S, Triponez F. Parathyroid gland angiography with indocyanine green fluorescence to predict parathyroid function after thyroid surgery. Br J Surg. 2016 Apr;103(5):537-43. doi: 10.1002/bjs.10101. Epub 2016 Feb 11. PMID 26864909
- [Background] Bergenfelz A, Barczynski M, Heie A, Muth A, Passler C, Schneider M, Wierzbicka P, Konturek A, Brauckhoff K, Elf AK, Dahlberg J, Hermann M. Impact of autofluorescence for detection of parathyroid glands during thyroidectomy on postoperative parathyroid hormone levels: parallel multicentre randomized clinical trial. Br J Surg. 2023 Nov 9;110(12):1824-1833. doi: 10.1093/bjs/znad278. PMID 37758507
- [Background] Benmiloud F, Godiris-Petit G, Gras R, Gillot JC, Turrin N, Penaranda G, Noullet S, Chereau N, Gaudart J, Chiche L, Rebaudet S. Association of Autofluorescence-Based Detection of the Parathyroid Glands During Total Thyroidectomy With Postoperative Hypocalcemia Risk: Results of the PARAFLUO Multicenter Randomized Clinical Trial. JAMA Surg. 2020 Feb 1;155(2):106-112. doi: 10.1001/jamasurg.2019.4613. PMID 31693081
- [Background] Thomas G, Squires MH, Metcalf T, Mahadevan-Jansen A, Phay JE. Imaging or Fiber Probe-Based Approach? Assessing Different Methods to Detect Near Infrared Autofluorescence for Intraoperative Parathyroid Identification. J Am Coll Surg. 2019 Dec;229(6):596-608.e3. doi: 10.1016/j.jamcollsurg.2019.09.003. Epub 2019 Sep 25. PMID 31562910
- [Background] Thomas G, McWade MA, Nguyen JQ, Sanders ME, Broome JT, Baregamian N, Solorzano CC, Mahadevan-Jansen A. Innovative surgical guidance for label-free real-time parathyroid identification. Surgery. 2019 Jan;165(1):114-123. doi: 10.1016/j.surg.2018.04.079. Epub 2018 Nov 12. PMID 30442424
- [Background] Thomas G, McWade MA, Paras C, Mannoh EA, Sanders ME, White LM, Broome JT, Phay JE, Baregamian N, Solorzano CC, Mahadevan-Jansen A. Developing a Clinical Prototype to Guide Surgeons for Intraoperative Label-Free Identification of Parathyroid Glands in Real Time. Thyroid. 2018 Nov;28(11):1517-1531. doi: 10.1089/thy.2017.0716. Epub 2018 Sep 11. PMID 30084742
- [Background] Paras C, Keller M, White L, Phay J, Mahadevan-Jansen A. Near-infrared autofluorescence for the detection of parathyroid glands. J Biomed Opt. 2011 Jun;16(6):067012. doi: 10.1117/1.3583571. PMID 21721833